CLINICAL TRIAL: NCT03810846
Title: Feasibility and Safety of Walking Football in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Federação Portuguesa de Futebol, Portugal (Unknown); Administração Regional de Saúde do Norte, Portugal (Other); Fédération Internationale de Football Association (Unknown)
Responsible Party: Principal Investigator, Romeu Mendes, Researcher, Universidade do Porto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISPUP-RMFIFA2018
Record Dates: First submitted 2019-01-10; First posted 2019-01-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Exercise; Physical Activity; Football; Walking Football; Type 2 Diabetes; Primary Health Care; Feasibility; Safety
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): Walking football exercise program
  Interventions: Behavioral: Walking football exercise program

INTERVENTIONS:
Behavioral: Walking football exercise program — Participants will be organized in two teams of 20 players. Each team will have 60-min walking football exercise sessions three times per week (non-consecutive days), during three months (36 sessions). Different walking football exercise strategies will be developed according to participants' motor skills and tested with dose-escalated intensity for its safety and enjoyment. Exercise intensity will range between light to vigorous. No submaximal or maximal exercises will be tested. Exercise sessions will be conducted on a sports hall (indoor court) by a football coach and supervised by an exercise physiologist and a nurse.

SUMMARY:
Our main challenge is to develop a novel physical activity intervention to promote exercise participation sustainability and effective health benefits in type 2 diabetes (T2D) population with minimum health risks. The relevance of this study is supported by four cornerstones: 1) The Portuguese love football and there seems to be a major potential in the implementation of football practice as part of the prevention and treatment of noncommunicable diseases for the middle-aged and elderly Portuguese population; 2) no studies have assessed the feasibility and safety of a walking football exercise program for middle-age and older patients with T2D; 3) the proposed investigation relies on robust methodology; 4) this intervention can have further sustainability with the enrollment of football clubs and primary health care units.

DETAILED DESCRIPTION:
This work will be a quasi-experimental study where we aim to test the feasibility and safety of walking football in patients with T2D. The recruitment of participants will be held in primary health care units by Family Medicine medical doctors. All participants will receive instructions to maintain daily-life routines (lifestyle-related physical activity and dietary pattern), and to continue with usual care (diabetes consultations on primary health care units and pharmacological regimen) along the studies duration. All participants will receive basic sports material (sports bag, T-shirt, and sports shoes). Participants will be organized in two teams of 20 players. Each team will have 60-min walking football exercise sessions three times per week (non-consecutive days), during three months (36 sessions). Different walking football exercise strategies will be developed according to participants' motor skills and tested with dose-escalated intensity for its safety (acute effects on capillary glycaemia, blood pressure, foot impact, exercise-related injuries and adverse events) and enjoyment. Exercise intensity will range between light to vigorous. No submaximal or maximal exercises will be tested. Cumulative short-term effects will also be analyzed along the three months through pre- and post-study evaluations. Exercise sessions will be conducted on a sports hall (indoor court) by a football coach and supervised by an exercise physiologist and a nurse.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of type 2 diabetes for at least 12 months;
* glycated hemoglobin bellow 10 %;
* not having started insulin therapy in the previous six months;
* not having started therapy with sulfonylureas in the previous six months;
* major complications of diabetes screened and controlled (diabetic retinopathy, diabetic nephropathy and diabetic foot);
* no symptoms of coronary artery disease;
* no cardiovascular, respiratory and musculoskeletal contraindications to exercise;
* not under cancer treatment (radiotherapy or intravenous chemotherapy);
* without limitations in gait or balance;
* independent living in the community;
* not engaged in supervised exercise;
* non-smokers at least for 6 months.

Exclusion Criteria:

* cardiological stress test with cardiac or hemodynamic problems

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Exercise intensity - subjective internal load | Through 3 months
  OMNI rating of perceived exertion scale during exercise (0 [lowest] to 10 [highest] points)
Exercise intensity - objective internal load | Through 3 months
  Heart rate during exercise
Exercise intensity - external load | Through 3 months
  Distance (km) assessed using GPS tracking during exercise
Acute glycemic effect | Change between before and immediately after each exercise session
  Acute change in capillary blood glucose with exercise sessions
Acute systolic blood pressure effect | Change between before and immediately after each exercise session
  Acute change in systolic blood pressure with exercise sessions
Acute diastolic blood pressure effect | Change between before and immediately after each exercise session
  Acute change in diastolic blood pressure with exercise sessions
Incidence of falls | Through 3 months
  Number of falls during the exercise program
Incidence of foot injuries | Through 3 months
  Number of reported foot injuries during the exercise program
Incidence of musculoskeletal injuries | Through 3 months
  Number of reported musculoskeletal injuries during the exercise program
Rate of Enjoyment | Through 3 months
  Self-reported exercise sessions' enjoyment on a likert scale (1 [lowest] to 5 [highest] points)

SECONDARY OUTCOMES:
Glycemic control | Change from baseline to 3 months
  Glycated hemoglobin (venous blood analysis)
Blood lipid profile | Change from baseline to 3 months
  Total cholesterol (venous blood analysis)
Clinical systolic blood pressure | Change from baseline to 3 months
  Resting systolic blood pressure
Clinical diastolic blood pressure | Change from baseline to 3 months
  Resting diastolic blood pressure
Body mass index | Change from baseline to 3 months
  Body mass index
Waist circumference | Change from baseline to 3 months
  Waist circumference
Body fat | Change from baseline to 3 months
  Body fat (bioelectrical impedance analysis)
Body lean mass | Change from baseline to 3 months
  Body lean mass (bioelectrical impedance analysis)
Agility/balance | Change from baseline to 3 months
  Timed Up and Go Test
Habitual physical activity | Change from baseline to 3 months
  Global Physical Activity Questionnaire
Food pattern | Change from baseline to 3 months
  24h-food recall analysis
Cognitive state | Change from baseline to 3 months
  Montreal Cognitive Assessment score (0 [lowest] to 30 [highest] points)
Health-related quality of life | Change from baseline to 3 months
  EQ-5D-5L questionnaire score (0 [lowest] to 100 [highest] points)
Medication | Change from baseline to 3 months
  Number of medications

CONTACTS AND LOCATIONS:
Overall Officials: Romeu Mendes, MD, PhD, Principal Investigator — EPIUnit - Instituto de Saúde Pública, Universidade do Porto
Locations (1):
- Instituto de Saúde Pública da Universidade do Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barbosa A, Brito J, Costa J, Ramos E, Firmino-Machado J, Seabra A, Figueiredo P, Sá MJ, Lunet N, Mendes R. SWEET-FOOTBALL: Development of an evidence-based walking football program for middle-aged and older patients with type 2 diabetes. Football is Medicine Conference 2019 - Programme and Abstracts. Odense: University of Southern Denmark; 2019. p. 32.
- [Result] Barbosa A, Brito J, Sá MJ, Puga F, Firmino-Machado J, Seabra A, Figueiredo P, Ramos E, Lunet N, Mendes R. Adherence and enjoyment of a walking-football program for patients with type 2 diabetes: SWEET-FOOTBALL Project. In: Bunc V, Tsolakidis E, editors. Book of Abstracts of the 24th Annual Congress of the European College of Sport Science. Prague: ECSS; 2019. p. 120-1.
- [Result] Rago V, Brito J, Costa J, Barbosa A, Figueiredo P, Seabra A, Travassos B, Mendes R. Activity profile during walking football training sessions in patients with type 2 diabetes. Football is Medicine Conference 2019 - Programme and Abstracts. Odense: University of Southern University; 2019. p. 41.
- [Result] Costa J, Brito J, Barbosa A, Figueiredo P, Seabra A, Sá MJ, Firmino-Machado J, Ramos E, Mendes R. Nocturnal cardiac autonomic activity in patients with type 2 diabetes engaged in a walking football programme. Football is Medicine Conference 2019 - Programme and Abstracts. Odense: University of Southern Denmark; 2019. p. 39.
- [Derived] Barbosa A, Brito J, Costa J, Figueiredo P, Seabra A, Mendes R. Feasibility and safety of a walking football program in middle-aged and older men with type 2 diabetes. Prog Cardiovasc Dis. 2020 Nov-Dec;63(6):786-791. doi: 10.1016/j.pcad.2020.06.014. Epub 2020 Jul 4. PMID 32634461